CLINICAL TRIAL: NCT04852562
Title: The Effect of Modified Radical Endoscopic Sinus Surgery on Chinese Patients With Eosinopilic Nasal Polyps
Brief Title: The Effect of Modified Radical Endoscopic Sinus Surgery on Eosinopilic Chronic Rhinosinusitus With Nasal Polyps
Acronym: EMRESSECRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zheng Liu (Other)
Collaborators: Wuhan Central Hospital (Other); Wuhan No.1 Hospital (Other); Tianyou Hospital Affiliated to Wuhan University of Science and Technology (Other); Wuhan Third Hospital (Other); Wuhan Pu-Ai Hospital (Other)
Responsible Party: Sponsor-Investigator, Zheng Liu, Professor of Otolaryngology-Head & Neck Surgery Vice Director Department of ENT Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENTmodifiedRESS-01
Record Dates: First submitted 2020-09-20; First posted 2021-04-21 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Chronic Sinusitis; Endoscopic Sinus Surgery; Nasal Polyps
Keywords: eosinophilic chronic rhinosinusitus with nasal polyps.; endoscopic sinus surgery; Nasal Polyps
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modified radical endoscopic sinus surgery(MRESS) (Experimental): The experimental group intends to adopt a modified radical endoscopic sinus surger to remove the mucosa including ethmoid sinus and maxillary sinus, as well as a completly middle turbinate resection to achieve a radical cure of ethmoid sinus. Antrostomies of frontal and sphenoid sinuses were then performed with meticulous operation and preserve the mucosa intactly.
  Interventions: Procedure: Modified radical endoscopic sinus surgery
- Functional endoscopic sinus surgery (FESS) (Experimental): FESS was performed by Messerklinger technique, operation procedures including full maxillary antrostomy, ethmoidectomy, sphenoidotomy and frontal sinusotomy, but with the middle turbinate preservation.
  Interventions: Procedure: functional endoscopic sinus surgery

INTERVENTIONS:
Procedure: Modified radical endoscopic sinus surgery — Modified radical endoscopic sinus surgery was performed to remove the mucosa including ethmoid sinus and maxillary sinus, as well as a completly middle turbinate.
  Other Names: MRESS
  Arms: Modified radical endoscopic sinus surgery(MRESS)
Procedure: functional endoscopic sinus surgery — Full maxillary antrostomy, ethmoidectomy, sphenoidotomy and frontal sinusotomy, but with the middle turbinate preservation.
  Other Names: FESS
  Arms: Functional endoscopic sinus surgery (FESS)

SUMMARY:
Functional endoscopic sinus surgery (FESS) is the pimary surgical treatment of CRS, characterized with the preservation of nasal structure and function.But the control of disease by surgery has been unsatisfactory. Recent studies have shown that patients with recurrent CRSwNP (usually with severe eosinophilic inflammation), more radical surgery may be more effective. The purpose of this prospective and randomized study is to determine the effect of endoscopic sinus surgery for extensive mucosal removal in patients with eosinophilic chronic rhinosinusitus with nasal polyps.

DETAILED DESCRIPTION:
Chronic rhinosinusitis with nasal polyps (CRSwNP) is a multifactorial inflammatory disorder that causes various symptoms including nasal obstruction, rhinorrhea, olfactory dysfunction, facial pain, and headache. Patients with significant eosinophilic inflammation usually accompanied with a higher recurrence rate and more severe clinical symptoms. Endoscopic sinus surgery (ESS) is recommended to patients who do not response well to conservative treatments. A retrospective study showed that postoperative polyp recurrence rate of patients with severe eosinophilic inflammation was significantly reduced by rebooting sinus mucosa. In this study, the experimental group intends to adopt a modified radical surger to remove the mucosa including ethmoid sinus and maxillary sinus, as well as a completly middle turbinate resection to achieve a extensive treatment of ethmoid sinus. Antrostomies of frontal and sphenoid sinuses were then performed with meticulous operation and preserve the mucosa intactly.

ELIGIBILITY:
Inclusion Criteria:

* CRSwNP is diagnosed according to EPOS clinical guidelines and met surgical requirements, the blood eosinophil count was greater than 0.22;
* Subjects/legal authorized representatives must understand the purpose and procedures of the study and voluntarily sign the informed consent, voluntarily participate in the study and comply with the study regulations, understand and comply with follow-up plan, and can correctly record the scale score, the administration frequency, accompanying drug use and adverse events, etc;
* The examinee must be 18-65 years old, male or non pregnant female, limited to Chinese;
* During the treatment and follow-up period, female subjects have no pregnancy and lactation plans;
* The subjects did not participate in other clinical trials in the past three months and agreed not to participate in other clinical trials before reaching the end point of this trial;
* Patients accompanying asthma must use their regular asthma treatment steadily in the past 6 weeks;

Exclusion Criteria:

* Women must not be pregnant, or breast-feeding;
* Subjects with cystic fibrosis, congenital ciliary dyskinesia, fungal sinusitis, systemic vasculitis and granulomatous disease, tumor, and immunodeficiency are exclued;
* Subjects accpted nasal endoscopic surgery within 6 months are exclued;
* Subjects with an upper respiratory tract infection within 4 weeks of entering the study are excluded;
* Subjects with serious metabolic, cardiovascular, autoimmune, neurology, blood, digestive, cerebrovascular, or respiratory system disease, or any disease interfering with the evaluation of results or affecting subjects safety are excluded, such as glaucoma and tuberculosis;
* Currently participating in other clinical studies or in other clinical investigators within 30 days, or staff directly involved in this study;
* Subjects with emotional or mental problems are excluded;
* Subjects must not have received immunotherapy within the previous 3 months;
* Subjects unsuitable for inclusion based on judgement of researchers are excluded;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-12-06 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline at months 1, 3, 6 and 12 in 22-item sino-nasaloutcome test (SNOT-22) scores after surgical intervention | 1month, 3month, 6month, 12month
  The SNOT-22 is a validated questionnaire that was used to assess the impact of chronic rhinosinusitis on health-related quality of life (HRQoL). It is a 22 item questionnaire with each item assigned a score ranging from 0 (no problem) to 5 (problem as bad as it can be). The total score may range from 0 (no disease) to 110 (worst disease), lower scores representing better health related quality of life.

SECONDARY OUTCOMES:
Revision surgery rate | 12month
  The rate of reoperation in each group after surgery
Symptom duration | 1month, 3month, 6month, 12month
  The time of duration of major symptoms of postoperative patients
Postoperative medication | 1month, 3month, 6month, 12month
  The duration and dose of postoperative medication needed to relieve symptoms
Recurrence time | 1month, 3month, 6month, 12month
  Recurrence was defined if the patient had symptoms of chronic rhinosinusitis after surgery, and nasal endoscopy found nasal polyps recurrence, obvious edema of mucosa, or purulent secretion, and above of symptoms or physical signs existed, which can't be alleviated by maximum medicine treatment at least 1 month
Change from baseline at months 1, 3, 6 and 12 in visual analogue scale (VAS) after surgical intervention | 1month, 3month, 6month, 12month
  The VAS for rhinosinusitis was used to evaluate the total disease severity. The participants were asked to indicate on a 10 centimeters (cm) VAS the answer to the question, "How troublesome are your symptoms of your rhinosinusitis?" The range of the VAS was from 0 (not troublesome) to 10 (worse thinkable troublesome), where higher score indicated worse thinkable troublesome.
Change from baseline at months 1, 3, 6 and 12 in nasal endoscopic score after surgical intervention | 1month, 3month, 6month, 12month
  Endoscopic result is scored according to Lund-Kennedy system, with the assessment of nasal polyp (NP), edema, nasal discharge, scarring and crusting. Items including edema, nasal discharge, scarring and crusting score 0 for no problem, 1 for mild abnormalities and 2 for severe abnormalities. NP score is graded and based on NP size recorded as the sum of the right and left nostril scores with a range of 0-8; higher scores indicate worse status. Individual score ranges from 0 (no polyps) to 4 (large polyps causing almost complete congestion/ obstruction of the inferior meatus) within each nostril.

OTHER OUTCOMES:
Changes from baseline at months 1, 3, 6 and 12 in molecular indices of nasal lavage fluid | 1month, 3month, 6month, 12month
  Investigate the change of inflammation molecular biomarkers using sample of nasal lavage fluid or mucosal lesion tissue. Biomarkers including interleukin 9, monocyte chemoattractant protein-1, macrophage inflammatory protein-1β, macrophage inflammatory protein-1α, chemokine (C-C motif ) ligand 17 and IgE in nasal lavage fluid at months 1, 3, 6 and 12 were detected to compare the changes of molecular indices relative to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Liu, Doctor, Study Chair — Huazhong University of Science and Technology
Locations (1):
- Department of ENT, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No